CLINICAL TRIAL: NCT02788591
Title: Confocal Endomicroscopy for Non-Erosive Reflux Disease Detection (CENERDD)
Brief Title: Confocal Endomicroscopy for Non-Erosive Reflux Disease Detection
Acronym: CENERDD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of accrual
Sponsor: LCMC Health (Other)
Responsible Party: Principal Investigator, Virendra Joshi, Physician, Gastroenterology, LCMC Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CENERDD
Record Dates: First submitted 2016-03-17; First posted 2016-06-02 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2021-10

CONDITIONS: Non-erosive Reflux Disease; Gastroesophageal Reflux
MeSH Terms: conditions — Non-Erosive Reflux Disease; Gastroesophageal Reflux | interventions — Proton Pump Inhibitors; Therapeutics; Omeprazole; Esomeprazole; Pantoprazole; Lansoprazole; Sucralfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proton Pump Inhibitor (PPI) Therapy (Other): 2x daily Proton Pump Inhibitor (PPI) Therapy for 8 weeks
  Interventions: Drug: Proton Pump Inhibitor (PPI) Therapy
- Sucralfate (Other): 4x daily Sucralfate slurry, 1g, for 8 weeks
  Interventions: Drug: Sucralfate

INTERVENTIONS:
Drug: Proton Pump Inhibitor (PPI) Therapy — Subject will take a proton pump inhibitor (PPI) of their choice (Omeprazole, Esomeprazole, Pantoprazole, or Lansoprazole) 2 times a day for 8 weeks.
  Other Names: Omeprazole, Esomeprazole, Pantoprazole, Lansoprazole
  Arms: Proton Pump Inhibitor (PPI) Therapy
Drug: Sucralfate — Subject will take Sucralfate 4 times a day for 8 weeks.
  Other Names: Carafate
  Arms: Sucralfate

SUMMARY:
Primary Objective:

Evaluate response to NERD treatment between patients with normal endomicroscopy findings compared with patients with abnormal endomicroscopy findings.

Secondary Objectives:

To evaluate the role of probe based endomicroscopy in the diagnosis of NERD by evaluating dilated intercellular spaces, evaluation of IPCL, and quantification of fluorescein leak.

Quality of life at study entry and end of study. Compare two medications under study within each group as a subgroup analysis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate response to non-erosive reflux disease (NERD) treatment between patients with normal endomicroscopy findings compared with patients with abnormal endomicroscopy findings. The researchers will compare two different drug regimens for the NERD subjects to evaluate their effectiveness in reducing NERD-related symptoms. In addition, the researchers will be testing the function and effectiveness of the confocal endomicroscopy procedure to be used during the study. Researchers will be continuing to assess the status, symptoms, and any changes associated with the symptoms subjects are experiencing.

The confocal endomicroscopy procedure utilizes a powerful microscope that is used during an endoscopy. An endoscopy is a procedure that allows us to scope/view the inside of the esophagus and stomach using a camera in precise detail.

An endoscopy procedure and measurements of acid in the esophagus have been used to determine if the investigators think acid is causing the symptoms. Traditionally, acid blocking medications called proton pump inhibitors (PPIs such as Esomeprazole, Lansoprazole, Omeprazole, and Pantoprazole), or medications such as Sucralfate have been used to treat the symptoms of NERD.

The medical community believes that these symptoms are due to increased spaces between the cells that make up the esophagus. They can directly see those spaces using the confocal endomicroscopy.

Patients are asked to participate in this study if they are 18 years of age or older and have typical symptoms for patients diagnosed with NERD that have not responded to the first attempted medication.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals older than 18 years who score a 12 or greater on the Reflux Disease Questionnaire and have failed a four week trial of daily proton pump inhibitor.
2. Subjects without gastroesophageal reflux disease (GERD) undergoing upper endomicroscopy for other indications will be recruited into study as controls.

Exclusion Criteria:

1. Barrett's esophagus
2. Use of twice daily proton pump inhibitor within 4 weeks of study entry
3. Esophageal varices
4. Coagulopathy (aspirin, NSAIDS and Plavix are allowed. Coumadin, Xarelto, heparin are not allowed.)
5. Gastrointestinal cancer or mass
6. Previous surgery involving the esophagus, stomach or duodenum
7. Pregnancy
8. Allergy to either sucralfate or proton pump inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Evaluate non erosive reflux disease (NERD) Symptoms. | 20 weeks
  Reflux Disease Questionnaire (RDQ)

SECONDARY OUTCOMES:
Evaluate the role of probe based endomicroscopy in the diagnosis of NERD by evaluating dilated intercellular spaces, evaluation of IPCL, and quantification of fluorescein leak. | 20 weeks
  A 3 minute video recording of microscopic images starting with the injection of the fluorescein will be captured during the time of endoscopy. The goal is also to see if the time to seeing fluorescein in the intracellular spaces correlates with a diagnosis of NERD. Time, measured in seconds, to first visualization of intrapapillary loops and intercellular gaps and fluorescein leak will be obtained and assess by trained endoscopists.
Compare quality of life in patients with NERD. | 20 weeks
  Quality of life questionnaire (SF-36)
Compare two medications within each NERD study groups as a subgroup analysis. | 20 weeks
  Categorical and binary demographics and outcomes will be assessed through a likelihood-ratio chi square test or a Fischer's exact test.Continuous outcomes, including time to fluorescein intracellular, will be assessed through a Student's t test or Wilcoxon rank sum, if the distribution of particular continuous variables is non-normal, tested through a Shapiro-Wilk statistic. Statistical significance will be determined at p values less than 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Joshi, MD, Principal Investigator — LCMC Health
Locations (2):
- United States (2):
  - Touro Infirmary New Orleans, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided